CLINICAL TRIAL: NCT05142930
Title: The Effect of Therapeutic Ultrasound on Pain in Coccydynia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Emel Güler, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02/29
Record Dates: First submitted 2021-11-16; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Coccyx Disorder
Keywords: coccyx; pain; ultrasonic waves
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Parallel groups will be received different treatment modalities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent ultrasound (Active Comparator): Patients with coccydynia will receive 10 sessions of physical therapy, 5 days a week for 2 weeks. Intermittent ultrasound will be used as a physical therapy agent. Intermittent ultrasound treatment will be applied to the muscles of the bilateral coccyx region at a dose of 1.0W/cm², at a frequency of 1 Megahertz, for 3+3 minutes.
  Interventions: Other: Intermittent ultrasound
- Continuous ultrasound (Active Comparator): Patients with coccydynia will receive 10 sessions of physical therapy, 5 days a week for 2 weeks. Continuous ultrasound will be used as a physical therapy agent. Continuous ultrasound treatment will be applied to the muscles of the bilateral coccyx region at a dose of 1.0W/cm², at a frequency of 1 Megahertz, for 3+3 minutes.
  Interventions: Other: Continuous ultrasound

INTERVENTIONS:
Other: Intermittent ultrasound — Intermittent ultrasound treatment will be applied to the muscles of the bilateral coccyx region
  Arms: Intermittent ultrasound
Other: Continuous ultrasound — Continuous ultrasound treatment will be applied to the muscles of the bilateral coccyx region
  Arms: Continuous ultrasound

SUMMARY:
Pain of the sacrococcygeal region is called coccydynia This painful clinical picture, which causes a decrease in the quality of life, also causes disability. Physical therapy modalities are used in the treatment of coccydynia. Ultrasound, which is used for diagnostic and therapeutic purposes, can be applied in two ways as continuous and intermittent for therapeutic purposes.Our aim in this study is to compare the effectiveness of continuous and intermittent ultrasound in patients with a diagnosis of coccydynia and to examine its effect on pain.

DETAILED DESCRIPTION:
Coccygodynia often develops from an inappropriate sitting position or when standing up from a sitting position. In the advanced stages of coccydynia, the pain becomes continuous. Conservative treatment, interventional procedures and surgical treatment are used in treatment. Medical treatment, physical therapy and local injection applications are accepted as conservative treatment methods.Among the physical therapy modalities, ultrasound has been used for many years in diseases affecting the musculoskeletal system. Ultrasound, which is used for diagnostic and therapeutic purposes, can be applied in two ways as continuous and intermittent for therapeutic purposes.

A total of 52 patients who applied between 01/04/2021 and 01/04/2022 and met the inclusion and exclusion criteria will be included in the study. Continuous ultrasound will be performed in 26 patients and intermittent ultrasound will be performed in 26 patients. Randomization will be determined by the treatment protocol prepared in closed envelopes.Within the scope of the study, the age, height, weight, trauma history, duration of complaint, severity of pain and Oswestry Disability Index scale will be recorded before the interventions. The patients will be followed up at the 3rd week and 3rd month after the treatment. The Oswestry Disability Index scale will be filled in to assess the severity of disability resulting from pain in the patient. Pain severity will be evaluated with the Visual Analog Scale (VAS).

Data will be entered into SPSS (version: 22.0) IBM SPSS statistical package program. Arithmetic mean, standard deviation, min-max, median values will be given in the data obtained by measurement. Percentage and frequency distribution will be given in the data obtained by counting. In statistical evaluations, parametric tests will be used for data showing normal distribution, and non-parametric tests will be used for data not showing normal distribution. Relationships will be compared according to the Pearson or Spearman correlation coefficient. Chi-square test will be applied to categorical data. P<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with coccydynia and having idiopathic or trauma history in etiology
* 18-75 years old
* The patient's acceptance of the ultrasound treatment to be applied
* Being in good mental health in terms of compliance with the treatment to be applied
* Receiving conservative treatment before ultrasound treatment
* The patient's numerical pain scale must be 5 and above

Exclusion Criteria:

* Being under the age of 18 and over the age of 75
* The patient's refusal to accept the treatment
* Wound or soft tissue infection in the skin area to be treated
* Pregnant patients
* Patients who have been diagnosed with malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | Change of VAS between baseline and at 3 weeks
  Visual Analog scale (VAS) will be used to determine the pain severity of patients.
Pain Severity | Change of VAS between baseline and at 3 months
  Visual Analog scale (VAS) will be used to determine the pain severity of patients.
Disability | Change of Owstery Disability Index between baseline and at 3 weeks
  Disability assessment will be made using the Owstery Disability Index. The scale consists of 10 items in total. Each item is graded between 0-5. As the total score increases, the level of disability increases. The maximum score is 50 points. The total score obtained from the patient will be converted into the percentage system and the disability percentage will be calculated and evaluated.
Disability | Change of Owstery Disability Index between baseline and at 3 months
  Disability assessment will be made using the Owstery Disability Index. The scale consists of 10 items in total. Each item is graded between 0-5. As the total score increases, the level of disability increases. The maximum score is 50 points. The total score obtained from the patient will be converted into the percentage system and the disability percentage will be calculated and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Emel Güler, MD, Principal Investigator — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haghighat S, Mashayekhi Asl M. Effects of Extracorporeal Shock Wave Therapy on Pain in Patients With Chronic Refractory Coccydynia: A Quasi-Experimental Study. Anesth Pain Med. 2016 Jun 1;6(4):e37428. doi: 10.5812/aapm.37428. eCollection 2016 Aug. PMID 27843777
- See also: Effect of extracorporeal shock wave therapy on coccydynia — http://pubmed.ncbi.nlm.nih.gov/27843777/